CLINICAL TRIAL: NCT01540175
Title: Immune Reconstitution in Oncology Patients Following Autologous Stem Cell Transplant
Acronym: IROPAST
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: XPD12-013 IROPAST
Record Dates: First submitted 2012-02-17; First posted 2012-02-28 (Estimated); Last update posted 2015-07-14 (Estimated); Status verified 2015-07

CONDITIONS: Solid Tumor; Brain Tumor; Lymphoma
Keywords: Autologous stem cell transplant; Immune reconstitution
MeSH Terms: conditions — Brain Neoplasms; Lymphoma | interventions — Phlebotomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants: Participants enrolled on the study will have blood samples obtained.
  Interventions: Other: Blood samples obtained

INTERVENTIONS:
Other: Blood samples obtained — Research participants agree to have blood samples obtained at the time of diagnosis before any chemotherapy, if available, and prior to high dose chemotherapy regimen with autologous HSCT as well as on days 14, 21, 28, week 8 and months 3, 6, 12 and 18 after autologous HSCT. Research participants with high risk neuroblastoma may also agree to have blood samples taken before and twice in the recovery period (days 0, 7 and 15-18) of Induction chemotherapy courses one and four.
  Other Names: Venipuncture; Phlebotomy

SUMMARY:
Autologous stem cell rescue is an established therapy in high risk neuroblastoma and relapsed Hodgkin's lymphoma and an experimental therapy in some other solid and brain tumors to facilitate the use of very intense chemotherapy beyond bone marrow tolerance. It is usually tolerated with acceptable toxicity and graft failure is practically not existent. But whereas immune reconstitution in allogeneic hematopoietic stem cell transplantation (HSCT) setting is widely studied, the investigators have no comprehensive data available in the autologous setting regarding recovery of the innate and adaptive immune system. However, observations in patients with autoimmune disease undergoing autologous HSCT suggest not an exact recovery of the patient's pre-transplant immune system but some re-education during reconstitution of immune function.

Also, recent developments of cancer-directed immunotherapy with monoclonal antibodies and immunocytokines rely on activity of the patient's own immune system via complement-mediated or antibody-dependent cellular cytotoxicity. These novel therapies are given either with or shortly after conventional chemotherapy. To find the optimal time point for administration of immunotherapy, it is important to know how and when immune effector cells recover after conventional myelosuppressive and/or immunosuppressive chemotherapy which are used in Induction regimens.

Researchers at St. Jude Children's Research Hospital want to study the research participant's immune profile once prior and at multiple set time points after autologous stem cell infusion during the recovery process. In a subset of participants the investigators want to study the recovery of lymphocyte subsets and function after one course of conventional chemotherapy preceding the high dose chemotherapy and autologous stem cell transplant. That way the investigators hope to learn about the pace and order of recovery and the functional capacity of different compartments of the immune system during reconstitution.

DETAILED DESCRIPTION:
Primary Objective:

* To describe the immune reconstitution of T cell-, B cell- and natural killer (NK) cell- compartment in patients undergoing autologous stem cell transplant as part of their treatment for a malignancy.

The design for this study will be a prospective, longitudinal observational study. Immune reconstitution will be measured in the course of autologous stem cell transplant using serial blood samples analyzed for cell counts, immune cell phenotyping (demonstrating the expression of specific receptors on the cell surface) and functional lymphocyte assays. These blood samples will be obtained once prior and at defined time points after stem cell infusion either while the research participant is hospitalized or during the scheduled clinic visit.

Immune recovery from conventional chemotherapy will be measured using serial blood samples analyzed for cell counts, immune cell phenotyping, and NK cell functional assays. These blood samples will be obtained once prior and at defined time points after completion of courses #1 and #4 of Induction chemotherapy while the research participant is hospitalized or during the scheduled clinic visit.

ELIGIBILITY:
Inclusion Criteria:

* Patients with solid tumors, brain tumors or lymphoma regardless of previously received cancer related therapies who are enrolled on a study protocol or treatment plan that includes or will likely include autologous stem cell transplant.
* Patient age >0 to 21 years

Exclusion Criteria:

* Patient receiving an autologous transplant for a disease other than listed above.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants will have a diagnosis of solid tumor, brain tumor or lymphoma, be 21 years of age or younger, and be enrolled on a protocol likely to include autologous stem cell transplant.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2012-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change in the immune reconstitution of T cell, B cell, and NK cell compartment. | Days 0, 14, 21, 28, week 8, and months 3, 6, 12, and 18 related to stem cell infusion.
  The order and magnitude of recovery of the different subtypes of leukocytes will be summarized by descriptive statistics. The pattern of immune reconstitution will be evaluated using longitudinal approaches such as Mixed effect models or GEE approach and implement in SAS 9.2 using PROC MIXED or PROC GENMOD.
  In addition, NK cell number, receptor and ligand genotype and phenotype and functional capacity will be compared at specific time points (28 days, 8 weeks and 6 months post autologous transplant) to the baseline values using paired one sample signed rank test.

CONTACTS AND LOCATIONS:
Overall Officials: Aimee Talleur, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org